CLINICAL TRIAL: NCT07005765
Title: The Effects of Video-Based Stabilization Exercises on Pain, Functionality, Exercise Adherence, Kinesiophobia, and Qol in Individuals With NSCBP
Brief Title: Effect of Video-based Stabilization Exercises on Pain, Function, Adherence, Kinesiophobia & QoL in NSCBP Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serra Sürel (Other)
Responsible Party: Sponsor-Investigator, Serra Sürel, Master's Student and Principal Investigator, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSurel-Tez2025
Record Dates: First submitted 2025-05-23; First posted 2025-06-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Non Specific Chronic Low Back Pain; Exercise Therapy
Keywords: Chronic Low Back Pain; Core Exercise; Exercise Adherence

STUDY DESIGN:
Intervention Model Description: Participants with non-specific chronic low back pain will be randomly assigned into two parallel groups. One group will receive a 6-week home-based stabilization exercise program delivered via video instructions, while the other group will receive the same exercise program using illustrated printed brochures. Both groups will follow the intervention independently without crossover. The effectiveness of the interventions will be compared between groups after 6 weeks.
Who Masked: Participant
Masking Description: Participants will be blinded to their group assignment and will not know whether they receive video-based or brochure-based exercise instructions. However, investigators delivering the interventions will be aware of the assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-Based Exercise Group (Experimental): Participants receive stabilization exercises delivered via video for 6 weeks.
  Interventions: Behavioral: Video-Based Stabilization Exercise Program
- Brochure-Based Exercise Group (Experimental): Participants receive the same stabilization exercises through illustrated brochures for 6 weeks.
  Interventions: Behavioral: Brochure-Based Stabilization Exercise Program

INTERVENTIONS:
Behavioral: Video-Based Stabilization Exercise Program — Participants will follow a 6-week home exercise program focusing on stabilization exercises. The instructions and demonstrations will be delivered through video format, which participants can watch at their convenience. The program aims to improve pain, functionality, exercise adherence, kinesiophobia, and quality of life.
  Arms: Video-Based Exercise Group
Behavioral: Brochure-Based Stabilization Exercise Program — Participants will follow the same 6-week home exercise program using illustrated printed brochures that provide step-by-step instructions for stabilization exercises. This format allows participants to perform exercises independently. The program's effects on pain, functionality, exercise adherence, kinesiophobia, and quality of life will be evaluated.
  Arms: Brochure-Based Exercise Group

SUMMARY:
This randomized controlled study aims to evaluate the effectiveness of a 6-week home-based stabilization exercise program in individuals with non-specific chronic low back pain. Participants will be randomly assigned to two groups: one receiving exercise instruction via video-based content, and the other via a printed brochure with illustrated exercises. The effectiveness of the interventions will be assessed in terms of pain severity, functional status, exercise adherence, kinesiophobia, and quality of life.

DETAILED DESCRIPTION:
This study investigates the effectiveness of a 6-week home-based core stabilization exercise program in individuals with non-specific chronic low back pain (NSCLBP). The purpose is to compare two different delivery methods of the same exercise protocol: video-based versus illustrated brochure-based instructions. Stabilization exercises are commonly used in NSCLBP management; however, the mode of delivery in home settings can impact adherence and clinical outcomes.

A total of 42 participants with NSCLBP will be randomly assigned to either the video-based group or the brochure-based group. Both groups will follow the same exercise content, frequency, and duration. Outcomes will be assessed at baseline and after 6 weeks using standardized tools for pain (Visual Analog Scale), functional status ( Oswestry Disability Index), exercise adherence (Exercise Adherence Rating Scale), kinesiophobia (Tampa Scale), and quality of life (SF-36).

The findings will be contribute to the optimization of home exercise strategies for chronic low back pain management.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of non-specific chronic low back pain lasting 3 months or more

Age 18 years or older

Score of 4 or higher on the Roland-Morris Disability Questionnaire

Voluntary agreement to participate in the study

Exclusion Criteria:

Physiotherapy treatment for low back pain within the past 6 months

Pain radiating to the lower extremities

Pregnancy

History of spinal surgery

Presence of central or peripheral nervous system pathology (e.g., stroke)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia | Baseline and after 6 weeks of intervention
  Kinesiophobia will be assessed using the Tampa Scale for Kinesiophobia (TSK), a validated self-report questionnaire that evaluates fear of movement or re-injury. The scale consists of 17 items rated on a 4-point Likert scale. The total score varies between 17 and 68. Higher scores indicate greater levels of fear.

SECONDARY OUTCOMES:
Pain Intensity | Baseline and after 6 weeks
  Pain will be measured using the Visual Analog Scale (VAS), scored from 0 (no pain) to 10 (worst pain).
Functional Disability | Baseline and after 6 weeks
  Functional disability will be assessed using the Oswestry Disability Index (ODI). The lowest score is 0 and the highest score is 50. Higher scores reflect greater disability.
Change in Quality of Life | Baseline and after 6 weeks
  Quality of life will be assessed with the Short Form-36 (SF-36), which evaluates physical, emotional, and social well-being. The total score varies between 0 (lowest quality of life score) and 100 (highest quality of life score).
Exercise Adherence | At the end of the 6-week intervention
  Exercise adherence will be assessed through an Exercise Adherence Rating Scale (EARS). Scoring ranges from 0 to 64. Higher scores indicate greater compliance with exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Kalaycı, PhD, PT, Principal Investigator — Bahçeşehir University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Camlik Medical Center, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No